CLINICAL TRIAL: NCT02670863
Title: Safety and Efficacy of a New Term Infant Formula Supplemented With A Prebiotic: a Doubleblind, Randomized, Controlled Trial
Brief Title: Safety and Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 14.15.INF
Record Dates: First submitted 2016-01-20; First posted 2016-02-02 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Infant Term Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Infant Formula (Experimental): Experimental Infant Formula containing a prebiotic
  Interventions: Other: Experimental Infant Formula
- Standard Infant Formula (Active Comparator): Standard bovine milk-based term infant formula
  Interventions: Other: Standard Infant Formula

INTERVENTIONS:
Other: Experimental Infant Formula — Standard bovine milk-based term infant formula supplemented with a prebiotic, fed ad libitum
  Arms: Experimental Infant Formula
Other: Standard Infant Formula — Standard bovine milk-based term infant formula, fed ad libitum
  Arms: Standard Infant Formula

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the experimental formula supplemented with a prebiotic vs the control formula.

DETAILED DESCRIPTION:
Randomized, double-blind, controlled interventional clinical trial design. The purpose of this study is to evaluate the safety and efficacy of a new term infant formula supplemented with a prebiotic vs a standard infant formula fed for 150 days to healthy, term infants.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Infants whose parent(s)/LAR have reached the legal age of majority in the Philippines
* Infants whose parent(s)/LAR are willing and able to comply with study requirements
* Infants whose parent(s)/LAR are able to be contacted by telephone throughout the study
* Healthy term, singleton infant at birth
* Between 21 to 26 days post-natal age at enrollment visit
* Weight-for-length and head circumference-for-age z-scores >/= - 3 and </= +3 according to WHO Child Growth Standards
* Infants of parent(s)/LAR who have previously made the decision to formula feed their infant at the time of enrollment

Exclusion Criteria:

* Infants with conditions requiring infant feedings other than those specified in the protocol
* Infants receiving complementary foods or liquids
* Infants who have a medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results
* Infants who are presently receiving or have received medications that could interfere with the interpretation of study results
* Infants or infants whose parents/LAR cannot be expected to comply with the protocol or with study procedures

Ages: 21 Days to 26 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 239 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Growth | 150 days
  weight gain velocity
Stool Consistency Score | 150 days

SECONDARY OUTCOMES:
Weight | 150 days
  weight in grams
Average Daily Stool Frequency | 150 days
Fecal Microbiota | 150 days
Fecal Markers | 150 days
Adverse Events | 150 days

CONTACTS AND LOCATIONS:
Overall Officials: Elvira M Estorninos, MD, Principal Investigator — Asian Hospital and Medical Center
Locations (1):
- Asian Hospital and Medical Center, City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: Undecided